CLINICAL TRIAL: NCT00170898
Title: A 7-Day Multicenter Randomized Double-Blind, Double-Dummy Parallel Group Trial to Assess the Safety and Efficacy of 400 mg Lumiracoxib Once Daily Versus 500 mg Naproxen Twice Daily in Patients With Acute Musculoskeletal Pain Due to Uncomplicated Soft Tissue Injury
Brief Title: Safety and Efficacy of Lumiracoxib Versus Naproxen in Acute Musculoskeletal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189AGB02
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-06

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal pain; cyclooxygenase-2 inhibitors; lumiracoxib; naproxen
MeSH Terms: conditions — Musculoskeletal Pain | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study is designed to develop our understanding of the risk-benefit of using lumiracoxib in patients with acute musculoskeletal pain due to uncomplicated soft tissue injury.

ELIGIBILITY:
Inclusion Criteria

* Patients with acute musculoskeletal pain following an uncomplicated soft tissue injury (within the last 72 hours) which is expected to be self-limiting, requiring short-term treatment with a NSAID.
* Patients' acute musculoskeletal pain at baseline must be ≥ 50 mm on a 0 - 100 mm on a Visual Analogue Scale.
* Patients may have taken analgesic therapy following injury. However, the baseline pain intensity assessment should be taken: (i) 4 hours after the last dose of ≤ 400 mg ibuprofen, ≤ 1000 mg paracetamol, ≤ 600 mg aspirin or ≤ 2 tablets of other over-the-counter analgesic aspirin-based or paracetamol-based combination medications (ii) or 8 hours after the last dose of > 400 mg ibuprofen or ≤ 50 mg diclofenac

Exclusion Criteria

* Patients whose pain is due to an acute exacerbation of a chronic condition e.g. osteoarthritis, rheumatoid arthritis, systemic lupus erythematosus.
* Patients who have taken non-steroidal anti-inflammatory drugs in the previous 24 hours (other than aspirin, ibuprofen, diclofenac, as described above).

Other protocol-defined inclusion/ exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 419
Dates: Start 2004-11

PRIMARY OUTCOMES:
Decrease in sum of pain intensity difference scores over first 5 days of treatment

SECONDARY OUTCOMES:
Decrease in sum of pain intensity difference scores over 7 days of treatment; Improvement in how pts feel about their pain; Comparable perceived pain relief; Comparable treatment satisfaction
Safety and efficacy as compared to naproxen.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals UK Limited Novartis Pharmaceuticals UK Limited, Study Director — Novartis Pharmaceuticals UK Limited
Locations (1):
- For site information contact, Novartis Pharmaceuticals UK Limited, Frimley, United Kingdom

REFERENCES:
- [Derived] Kyle C, Zachariah J, Kinch H, Ellis G, Andrews C, Adekunle F. A randomised, double-blind study comparing lumiracoxib with naproxen for acute musculoskeletal pain. Int J Clin Pract. 2008 Nov;62(11):1684-92. doi: 10.1111/j.1742-1241.2008.01906.x. PMID 19143855